CLINICAL TRIAL: NCT01636284
Title: A Single-Arm, Open-Label Phase 2 Study of JX 594 (Thymidine Kinase-Deactivated Vaccinia Virus Plus GM-CSF) Administered by Weekly Intravenous (IV) Infusions in Sorafenib-naïve Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: A Phase 2a Study of Modified Vaccinia Virus to Treat Sorafenib-naïve Advanced Liver Cancer
Acronym: FLASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennerex Biotherapeutics (Industry)
Responsible Party: Sponsor
Organization: SillaJen, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JX594-IV-HEP021
Record Dates: First submitted 2012-06-23; First posted 2012-07-10 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Hepatocellular Carinoma
Keywords: Liver Cancer; HCC; first line HCC; Pexa-Vec; JX-594
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- JX-594 recombinant vaccina GM-CSF (Experimental): JX-594 recombinant vaccina GM-CSF
  Interventions: Biological: JX-594 recombinant vaccina GM-CSF

INTERVENTIONS:
Biological: JX-594 recombinant vaccina GM-CSF — Enrolled patients will receive 5 weekly IV infusions on Days 1, 8, 15, 22, and 29. After Day 43, if their disease has improved or remained stable and they have not started other cancer therapy, they may be able to continue to receive JX-594 via IV infusion every three weeks. This treatment extension may continue until radiologic progressive disease, initiation of other cancer therapy, or patient withdrawal.

SUMMARY:
This study is to determine how effectively JX-594 (Pexa-Vec) will prolong life in patients with advanced Hepatocellular Carcinoma (HCC) who have not been previously treated with sorafenib, and the safe administration of JX-594 in five weekly IV infusions.

DETAILED DESCRIPTION:
This was a Phase 2a, two-staged, single-arm, open-label study in sorafenib-naïve patients with advanced HCC.

Patients received 5 weekly IV infusions of Pexa-Vec and could have continued to receive IV infusions of Pexa-Vec every 3 weeks until progressive disease (PD).

ELIGIBILITY:
KEY Inclusion Criteria:

* Histologic or cytologic confirmation of advanced primary hepatocellular carcinoma (HCC)
* Measurable tumor (at least one tumor with ≥1 cm LD of contrast-enhancement during the arterial phase on CT scanning)
* ECOG performance status 0, 1 or 2
* Child-Pugh Class A; or Child-Pugh Class B7 without clinically significant ascites
* Platelet count ≥50,000 plts/mm3
* WBC count ≥2,000 cells/mm3 and ≤50,000 cells/mm3
* Hemoglobin ≥10 g/dL
* Adequate liver function

KEY Exclusion Criteria:

* Received sorafenib as previous treatment for HCC for more than 14 days
* History of severe exfoliative skin condition (e.g., eczema or atopic dermatitis requiring systemic therapy for > 4 weeks)
* Prior treatment with JX-594
* Known significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication
* Severe or unstable cardiac disease
* Viable CNS malignancy associated with clinical symptoms
* Pregnant or nursing an infant
* Significant bleeding event within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Burke, MD, Study Director — Jennerex Biotherapeutics
Locations (5):
- United States (2):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- South Korea (2):
  - Pusan National University Hospital, Pusan
  - Pusan National University Yangsan Hospital, Yangsan
- University Clinic of Navarra, Pamplona, Navarre, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | JX-594 Recombinant Vaccina GM-CSF
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | JX-594 Recombinant Vaccina GM-CSF
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 13
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Radiographic Response
Description: Number of Participants with Complete response [CR] or partial response [PR] per modified Response Evaluation Criteria in Solid Tumors (mRECIST) for target and non-target lesions assessed by enhanced CT scan: CR, disappearance of intratumoral enhancing area; PR, >=30% decrease in sum of diameters of enhancing area; Radiographic Response = CR + PR
Time Frame: CT scans every 6 week from Week 6 up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | JX-594 Recombinant Vaccina GM-CSF
Number analyzed (Participants) | 16
Participants | 4

2. Secondary Outcome: Time to Progression (TTP)
Description: TTP (in months) was defined as the number of months from the date of first Pexa-Vec infusion to the date of disease progression. If the patient had no progression then TTP was censored at the date of last evaluable tumor assessment. TTP was summarized and a Kaplan Meier (KM) curve was constructed.
Time Frame: CT scans every 6 week from Week 6 up to 12 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | JX-594 Recombinant Vaccina GM-CSF
Number analyzed (Participants) | 16
months | 1.38 [1.35 to 2.73]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of Pexa-Vec until death from any cause. For patients not known to have died at the time of the analysis, OS was censored on the date they were last known to be alive. OS was summarized and a KM curve was constructed.
Time Frame: CT scans every 6 week from Week 6 up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | JX-594 Recombinant Vaccina GM-CSF
Number analyzed (Participants) | 16
months | 7.47 [4.44 to 10.64]

ADVERSE EVENTS:
Time Frame: From the date when ICF signed up to 12 months
Arm/Group | JX-594 Recombinant Vaccina GM-CSF
All-Cause Mortality (participants affected / at risk) | 3/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JX-594 Recombinant Vaccina GM-CSF (N=16)
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Liver Carcinoma Ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Hepatorenal Syndrome (Hepatobiliary disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JX-594 Recombinant Vaccina GM-CSF (N=16)
Chills (General disorders) | 13
Influenza Like Illness (General disorders) | 13
Pyrexia (General disorders) | 9
Fatigue (General disorders) | 3
Oedema Peripheral (General disorders) | 3
Pain (General disorders) | 2
Chest Discomfort (General disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 5
Ascites (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Abdominal Distension (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 7
Rash Pustular (Infections and infestations) | 5
Upper Respiratory Tract Infection (Infections and infestations) | 3
Herpes Zoster (Infections and infestations) | 2
Acute Tonsillitis (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Decreased Appetite (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Aspartate Aminotransferase Increased (Investigations) | 4
Platelet Count Decreased (Investigations) | 3
Alanine Aminotransferase Increased (Investigations) | 2
Blood Bilirubin Increased (Investigations) | 1
Eosinophil Count Increased (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 1
Neutrophil Count Increased (Investigations) | 1
White Blood Cell Count Decreased (Investigations) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 2
Productive Cough (Musculoskeletal and connective tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Cold Sweat (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash Generalised (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 3
Tachycardia (Cardiac disorders) | 3
Jaundice (Hepatobiliary disorders) | 2
Hepatic Failure (Hepatobiliary disorders) | 1
Hepatorenal Syndrome (Hepatobiliary disorders) | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Liver Carcinoma Ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases To Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysuria (Renal and urinary disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Insomnia (Psychiatric disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No